CLINICAL TRIAL: NCT04139551
Title: Oxford Study of Quantification in Parkinsonism Study - OXQUIP
Brief Title: Oxford Study of Quantification in Parkinsonism
Acronym: OxQUIP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Oxford (Other)
Collaborators: UCB Belgium (Unknown)
Responsible Party: Sponsor
Other Study IDs: IRAS ID 211382; 16/SW/0262 REC reference (Other: University of Oxford)
Record Dates: First submitted 2019-10-18; First posted 2019-10-25 (Actual); Last update posted 2020-12-11 (Actual); Status verified 2020-08

CONDITIONS: Parkinson Disease; Progressive Supranuclear Palsy
Keywords: wearable technology; Saccadic eye movements; Gait assessment; Cognitive tests
MeSH Terms: conditions — Parkinson Disease; Supranuclear Palsy, Progressive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- 1XXX Denono PD: Newly diagnosed unmedicated PD patients
- 2XXX Mild /Moderate PD: Early to moderate stage PD patients well controlled on medication(typically fewer than 8 years since diagnosis)
- 3XXX Advanced PD: Advanced PD patients (typically greater than 8 years duration)
- 4XXX DBS patients: PD patients with deep brain stimulation systems
- 5XXX PSP patients: PSP patients
- 6XXX Healthy Controls: Age-frequency matched healthy controls

SUMMARY:
The OxQUIP (Oxford QUantification In Parkinsonism) study is recruiting patients with Parkinson's Disease and Progressive Supranuclear Palsy. Currently available treatments for these diseases are symptomatic only, and do not have any preventive or disease-slowing effect. As new drugs are developed, there is a need to be able to evaluate them quickly, so that precious time and resources can be devoted to those showing most promise.

This study follows participants intensively over an initially 3 year period, with the aim of identifying measures that can detect disease progression over much shorter time periods than is possible at present.

During the study participants are asked to perform simple tasks while the investigators measure movements of the eyes, hands and body. The investigators also do some tasks on a tablet computer that measure cognitive performance.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a common neurodegenerative disease that affects one in every hundred people over the age of 55. It is estimated that there are seven to ten million people with PD worldwide. It is disabling, incurable and gradually progressive. Progressive Supranuclear Palsy (PSP) is a related condition that presents initially with very similar features to PD. Eventually other features appear that are not part of idiopathic PD, such as paralysis of voluntary upgaze. Currently available treatments for both PD and PSP are symptomatic only, and while they may be effective for a number of years, they do not have any preventive or disease-slowing effect.

One of the problems with these conditions is that presently, there is a lack of completely reliable means of measuring their severity. The investigators use "clinical rating scales" which are points-based systems in which a doctor or nurse has to score how badly the person with PD or PSP is affected by various aspects of their condition. This is a subjective process, in other words it depends on the impression of the person making the assessment, and two doctors may sometimes disagree about the score. The scale is also sometimes difficult to interpret, for example the difference between scores of 20 and 30 may not be the same size as the difference between scores of 30 and 40. In contrast, most medical conditions nowadays can be very accurately and reliably measured using special equipment, for example the level of a patient's blood pressure, or the difficulty of breathing in asthma.

The need for accurate measures is particularly great when conducting trials of new drugs. Accurate evaluation of whether they work or not depends on precise measures of disease symptoms for each patient both before and after treatment. Drug trials may take years, and an accurate early measure of effect would allow interim results to guide decisions at which point resources can be focussed on those drugs that look most promising.

The aim of this study is to develop and validate sensitive tests to measure the symptoms of PD and PSP.

ELIGIBILITY:
Inclusion Criteria:

* The participant may enter the study as a patient participant if ALL of the following apply:

  * Participant is willing and able to give informed consent for participation in the study
  * Fluent in English
  * Male or Female, aged 50 years or above
  * Patient diagnosed with PD or PSP by a specialist movement disorders neurologist, or age matched healthy control (often but not always the spouse of a patient)
  * No evidence of significant cognitive impairment
  * Normal or corrected-to-normal vision in both eyes

The participant may enter the study as a healthy control if ALL of the following apply:

* Participant is willing and able to give informed consent for participation in the study
* Fluent in English
* Male or Female, aged 50 years or above
* No history of neurological disease
* No evidence of significant cognitive impairment
* Normal or corrected-to-normal vision in both eyes

Exclusion Criteria:

The participant may not enter the study if ANY of the following apply:

* Patient is unwilling or unable to give informed consent.
* Significant neurological co-morbidity that may obfuscate interpretation of neurophysiological or cognitive test results, for example major stroke.
* Severe mental impairment due to dementia or psychosis
* Medical or psychiatric illness that would interfere with completing initial or any of the follow up assessments
* History of photosensitive epilepsy

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Parkinson's and Progressive Supranuclear Palsy patients along with aged - matched healthy controls.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2016-10 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Saccadic eye movements | 3 months, 6 months, 12 months, 18 months, 21 months, 24 months, 27 months and 30 months.
  Automated measurements of rapid conjugate eye movements using a device called a saccadometer.
Hand tapping | 3 months, 6 months, 12 months, 18 months, 21 months, 24 months, 27 months and 30 months
  Measurement of rate of hand tapping movements made by participant on an electronic pad.
Reaction times using a button box | 3 months, 6 months, 12 months, 18 months, 21 months, 24 months, 27 months and 30 months
  Measurement of response time when participant is required to press a button when a light is illuminated.
Gait measurement | 3 months, 6 months, 12 months, 18 months, 21 months, 24 months, 27 months and 30 months
  Characterisation of gait abnormalities using a body-worn array of inertial measurement units
Mini Mental State Examination (MMSE) cognitive tablet | 3 months, 6 months, 12 months, 18 months, 21 months, 24 months, 27 months and 30 months
  This is a standard clinical test for cognitive impairment
Montreal Cognitive Assessment (MOCA) | 3 months, 6 months, 12 months, 18 months, 21 months, 24 months, 27 months and 30 months
  This is a standard clinical test for cognitive impairment
Verbal fluency test measurement | 3 months, 6 months, 12 months, 18 months, 21 months, 24 months, 27 months and 30 months
  Measures a participant's ability to produce a list of words according to set criteria e.g. words starting with a specific letter of the alphabet.
Executive function testing (Oxford Cognitive Screen) | 3 months, 6 months, 12 months, 18 months, 21 months, 24 months, 27 months and 30 months
  This is an electronic tablet-based battery of tasks intended to screen for deficits in executive function.

CONTACTS AND LOCATIONS:
Overall Officials: Chrystalina A Antoniades, Principal Investigator — University of Oxford
Locations (1):
- John Radcliffe Hospital, Headington, Please Select, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Via scientific publications and several collaborations that are already under way.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be available two years after publication for a period of 10 years.
Access Criteria: Anyone interested can get in touch with our team and we will assess each request on case by case

REFERENCES:
- [Result] Lu Z, Buchanan T, Kennard C, FitzGerald JJ, Antoniades CA. The effect of levodopa on saccades - Oxford Quantification in Parkinsonism study. Parkinsonism Relat Disord. 2019 Nov;68:49-56. doi: 10.1016/j.parkreldis.2019.09.029. Epub 2019 Sep 27. PMID 31621619
- [Result] Patel S, Fitzgerald JJ, Antoniades CA. Oculomotor effects of medical and surgical treatments of Parkinson's disease. Prog Brain Res. 2019;249:297-305. doi: 10.1016/bs.pbr.2019.04.020. Epub 2019 May 20. PMID 31325988
- [Result] De Vos M, Prince J, Buchanan T, FitzGerald JJ, Antoniades CA. Discriminating progressive supranuclear palsy from Parkinson's disease using wearable technology and machine learning. Gait Posture. 2020 Mar;77:257-263. doi: 10.1016/j.gaitpost.2020.02.007. Epub 2020 Feb 10. PMID 32078894
- See also: Group website — http://www.ndcn.ox.ac.uk/research/neurometrology-lab/